CLINICAL TRIAL: NCT00180414
Title: MODULA-Study: Modul 7 VRR: Correlation Between Ventricular Rate Regulation (VRR) and the Percentage of Biventricular Pacing as Well as Subjective Quality of Life and Level of Physical Ability in CRT Patients With Atrial Fibrillation
Brief Title: MODULA Modul 7 VRR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrolment rate
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Guidant Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version vom 10.07.2003 BIS
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2022-03-29 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Atrial Fibrillation
Keywords: heart failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Ventricular Rate Regulation feature ON (Experimental)
  Interventions: Device: CRT devices with ventricular rate regulation [VRR] (CE labeled)
- Ventricular Rate Regulation feature OFF (Active Comparator)
  Interventions: Device: CRT devices with ventricular rate regulation [VRR] (CE labeled)

INTERVENTIONS:
Device: CRT devices with ventricular rate regulation [VRR] (CE labeled)

SUMMARY:
This study will look at the correlation between ventricular rate regulation (VRR) and the percentage of biventricular pacing as well as subjective quality of life and level of physical ability in CRT patients with atrial fibrillation.

DETAILED DESCRIPTION:
To investigate whether VRR can increase the amount of biventricular pacing in CRT patients with conducted atrial arrhythmias. Secondarily, an investigation will be carried out to determine whether this increase in biventricular pacing results in an improvement in quality of life, as well as an improvement in the symptoms caused by the atrial arrhythmia and an improvement in the level of physical ability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CRT system with the VRR algorithm
* Patients with permanent atrial fibrillation
* Occasional conducted atrial fibrillation resulting in ventricular rates > 70 beats per minute (bpm)
* QRS complex > 120 ms

Exclusion Criteria:

* Patients with third degree atrioventricular (AV) block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-08-28 (Actual); Primary Completion 2008-05-07 (Actual); Study Completion 2008-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Lemke, MD, Principal Investigator — Klinikum Lüdenscheid / Kardiologie / Paulmannshöher Straße 14 / 58515 Lüdenscheid / Germany
Locations (1):
- Klinikum Lüdenscheid / Kardiologie, Lüdenscheid, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Ventricular Rate Regulation Feature ON; Ventricular Rate Regulation Feature OFF: CRT devices with ventricular rate regulation [VRR] (CE labeled)
Period: Overall Study
Arm/Group | Ventricular Rate Regulation Feature ON | Ventricular Rate Regulation Feature OFF
Started | 4 | 4
Completed | 0 | 0
Not Completed | 4 | 4
Not completed — Study cancellation due to lack of overall enrollments | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ventricular Rate Regulation Feature ON | Ventricular Rate Regulation Feature OFF | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Only aggregate data for total cohort from final report available. No data or analysis per group available from final report. Individual data deleted meanwhile per applicable data storage regulations and unavailable for further analysis, hence this data is impossible to be provided. | NA (NA) — Only aggregate data for total cohort from final report available. No data or analysis per group available from final report. Individual data deleted meanwhile per applicable data storage regulations and unavailable for further analysis, hence this data is impossible to be provided. | 72.3 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Biventricular Pacing
Description: Comparison of the average percentage of biventricular pacing in subjects randomised to Ventricular Rate Regulation (VRR) = ON to subjects randomized to VRR = OFF
Time Frame: 6 month
Population: An insufficient number of subjects was enrolled as well as the overall data quality of this investigation did not allow for any conclusions regarding the endpoint. Endpoints were not analyzed, final report does not contain information about analysis. Individual data deleted meanwhile per applicable data storage regulations and unavailable for further analysis, hence detailed results are impossible to be provided.
Arm/Group | Ventricular Rate Regulation Feature ON | Ventricular Rate Regulation Feature OFF
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Correlation Between VRR and the Subjective Quality of Life
Description: Correlation between VRR mode and the subjective quality of life (QOL) measured by a QOL questionnaire in both randomized groups
Time Frame: 6 Month
Population: as for outcome 1
Arm/Group | Ventricular Rate Regulation Feature ON | Ventricular Rate Regulation Feature OFF
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Correlation Between VRR and the Symptoms Caused by Conducted Atrial Arrhythmias
Description: Correlation between VRR mode and conducted atrial arrhythmias (if observed) in both randomized groups
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Ventricular Rate Regulation Feature ON | Ventricular Rate Regulation Feature OFF
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Correlation Between VRR and Physical Ability (6 Minute Walk Test, Optional Spiroergometry)
Description: Correlation between VRR and physical ability in both randomized groups measured by a 6 minute walk test or an optional spiroergometry
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Ventricular Rate Regulation Feature ON | Ventricular Rate Regulation Feature OFF
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ventricular Rate Regulation Feature ON | Ventricular Rate Regulation Feature OFF
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes